CLINICAL TRIAL: NCT00366418
Title: A Pilot Study of Fractionated Dose Subcutaneous Rituximab (RTX, Rituxan(Registered Trademark)) in Patients With Refractory or Relapsed Chronic Lymphocytic Leukemia
Brief Title: Lower But More Frequent Dose Rituximab to Treat Chronic Lymphocytic Leukemia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 060228; 06-H-0228; NCT00389961 (obsolete NCT alias)
Record Dates: First submitted 2006-08-17; First posted 2006-08-21 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2011-02-23

CONDITIONS: Refractory Chronic Lymphocytic Leukemia
Keywords: CLL; Monoclonal Antibody Therapy; Anti CD20; Biologic Response Modifier Therapy; Fractionated-Dose; Low-Dose; Chronic Lymphocytic Leukemia
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — Rituximab

INTERVENTIONS:
Drug: Rituximab

SUMMARY:
This study will test the safety and effectiveness of using lower-dose rituximab given more frequently for treating chronic lymphocytic leukemia (CLL). Studies have shown that, used once a week for 4 weeks, rituximab was effective in up to 25 percent of patients with CLL. New evidence shows that using lower and more frequent doses of rituximab can be more effective in destroying leukemia cells and produce a better treatment response.

Patients 21 years of age and older with CLL who have received treatment with fludarabine may be eligible for this study.

Participants take rituximab for 12 weeks. One dose of the drug is infused through an arm vein over about 30 minutes on either day 1 (the first dose) or day 3 (the second dose). All other doses are given as an injection under the skin. After the first week, patients can choose to do these injections at home. Rituximab will be given 3 times a week for a total of 12 weeks. Other medications are given to reduce the side effects and allergic reactions to the drug. In addition to treatment, patients undergo the following tests and procedures:

Before treatment

* Medical history, physical examination, electrocardiogram (EKG) and blood tests.
* Bone marrow and lymph node biopsies (surgical removal of a small tissue sample).
* Computed tomography (CT) and positron emission tomography (PET) scans. CT uses special x-rays to provide images of the neck, chest, abdomen and pelvis. PET uses a radioactive sugar to identify areas of disease.

During treatment (study weeks 1-12)

* Medical history and physical examinations at weeks 3, 6 and 12 to evaluate drug side effects, plus weekly telephone checks and interim visits when needed.
* Blood tests every other week to evaluate blood counts.

Evaluations after treatment (follow-up 3 months to 12 months)

* Blood tests at follow-up visits at 3, 6, 9 and 12 months after treatment to evaluate blood counts.
* Bone marrow aspiration and biopsy at 3 months after treatment to examine the effects of rituximab on bone marrow cells.
* CT scans of the neck, chest, abdomen and pelvis at 3, 6, 9 and 12 months after treatment to evaluate the response to treatment.

DETAILED DESCRIPTION:
Rituximab is FDA approved for the treatment of relapsed or refractory low grade or follicular CD20+ B cell non Hodgkin's lymphoma (375 mg/m(2) IV infusion once weekly for 4 or 8 doses). Recently, rituximab (anti CD20) has been introduced to CLL treatment regimens and has become an attractive choice in combination chemotherapy or as single agent treatment. Rituximab has been shown to be effective at lower doses than 375 mg/m(2) when given more frequently.

Several theoretical considerations and supporting laboratory evidence suggest that a fractionated dosing schedule using low-dose rituximab could be more effective than the current i.v. schedule of high-dose rituximab. Indeed, preliminary clinical evidence suggests that low-dose rituximab at 20mg/m2 i.v. 3-times per week can lead to steady clearance of leukemic cells without inducing substantial loss of targeted CD20.

This is a Phase I/II , single agent study which will evaluate the safety and feasibility of subcutaneous rituximab (Rituxan) administered at 20 mg/day three times a week for 12 weeks in subjects with CLL. Patients need to have had prior treatment with fludarabine, and have an elevated absolute lymphocyte count. The primary objective will be to test the safety and feasibility of giving rituximab subcutaneously. We will also obtain as a secondary endpoint an early estimate of efficacy as evidenced by (a) shrinkage of lymphadenopathy and/or (b) improvement in blood values and bone marrow biopsy findings.

ELIGIBILITY:
* INCLUSION CRITERIA
* Patients diagnosed with Chronic Lymphocytic Leukemia
* Prior therapy with fludarabine or a fludarabine containing regimen
* CD20 expression on CLL cells
* Neutrophil count ANC greater than 500/mm(3)
* Platelet count greater than 30K/mm(3)
* Age 21-99

EXCLUSION CRITERIA

* Bulky lymphadenopathy, defined as greater than 1 lymph node with greater than 5cm in largest diameter
* Evidence for transformation into high grade lymphoma (Richter's transformation)
* ECOG performance 3 or higher
* Other concurrent anticancer therapies
* Less than 3 months from last systemic therapy for CLL
* Less than 6 months from last monoclonal antibody therapy
* More than 10 doses rituximab, within 12 months preceeding protocol enrollment, either as single agent or in a combination chemotherapy regimen
* Chronic or current clinically significant infection, including HIV positivity or hepatitis C
* Moribund status or concurrent hepatic, renal, cardiac, neurologic, pulmonary, infectious, or metabolic disease of such severity that it would preclude the patient's ability to tolerate protocol therapy
* History of mucocutaneous reactions (paraneoplastic pemphigus, Stevens-Johnson syndrome, lichenoid dermatitis, vesiculobullous dermatitis, and toxic epidermal necrolysis)
* Known anaphylaxis or IgE mediated hypersensitivity to murine proteins or to any component of this product
* Inability to self inject the study medication or to have it administered by a third person
* Inability to understand the investigational nature of the study ability to provide informed consent

Ages: 21 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2006-08-10; Primary Completion 2009-06-11 (Actual); Study Completion 2009-06-11 (Actual)

PRIMARY OUTCOMES:
Safety profile and early evidence of efficacy of Rituxan given subcutaneously. | 12 weeks

SECONDARY OUTCOMES:
Measurement/deposition of serum compliment components, analysis of rituxan induced gene and protein expression in CLL cells, analysis and binding of rituximab to CLL cells. | 1-12 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Chiorazzi N, Rai KR, Ferrarini M. Chronic lymphocytic leukemia. N Engl J Med. 2005 Feb 24;352(8):804-15. doi: 10.1056/NEJMra041720. No abstract available. PMID 15728813
- [Background] Beum PV, Kennedy AD, Williams ME, Lindorfer MA, Taylor RP. The shaving reaction: rituximab/CD20 complexes are removed from mantle cell lymphoma and chronic lymphocytic leukemia cells by THP-1 monocytes. J Immunol. 2006 Feb 15;176(4):2600-9. doi: 10.4049/jimmunol.176.4.2600. PMID 16456022
- [Background] Kennedy AD, Beum PV, Solga MD, DiLillo DJ, Lindorfer MA, Hess CE, Densmore JJ, Williams ME, Taylor RP. Rituximab infusion promotes rapid complement depletion and acute CD20 loss in chronic lymphocytic leukemia. J Immunol. 2004 Mar 1;172(5):3280-8. doi: 10.4049/jimmunol.172.5.3280. PMID 14978136
- [Derived] Aue G, Lindorfer MA, Beum PV, Pawluczkowycz AW, Vire B, Hughes T, Taylor RP, Wiestner A. Fractionated subcutaneous rituximab is well-tolerated and preserves CD20 expression on tumor cells in patients with chronic lymphocytic leukemia. Haematologica. 2010 Feb;95(2):329-32. doi: 10.3324/haematol.2009.012484. Epub 2009 Aug 13. PMID 19679883